CLINICAL TRIAL: NCT03435198
Title: Biomarkers in Exhaled Breath of Glucose Fluctuation in Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: East Tennessee State University (Other)
Collaborators: Mountain States Health Alliance (Unknown)
Responsible Party: Principal Investigator, Evan Los, Assistant Professor, East Tennessee State University
Other Study IDs: 0817.5f
Record Dates: First submitted 2018-01-30; First posted 2018-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Volatile Organic Compounds; Hypoglycemia; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — human breath samples collected in sealed bags and shipped to receiving/processing lab. Once processed, samples are destroyed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Collect exhaled breath during low and normal blood sugar — Collect exhaled breath during low and normal blood sugar to determine if there are any differences between the two in people with type 1 diabetes.

SUMMARY:
The investigators are investigating the "biochemical fingerprint" of hypoglycemia (low blood sugar) in the breath of people with type 1 diabetes.

DETAILED DESCRIPTION:
The investigators aim through the use of proton-transfer-reaction mass spectrometry to perform comprehensive breath analysis to identify compounds of interest associated with glucose fluctuations. More than 500 different volatile organic compounds can be detected in human breath. Compounds such as ethane, pentane and isoprene (hydrocarbons), as well as acetone, acetaldehyde, methanol, ethanol, 2-propanol (oxygen-containing compounds), are most likely to be relevant and measurable in our study population. Hydrocarbons are stable end-products of lipid peroxidation and show only low solubility in blood and therefor are excreted into breath within minutes of their formation in tissues. There is evidence for increased hydrocarbon production in states of oxidative stress. Oxygen-containing compounds such as acetone/acetaldehyde (ketones) are also clinically relevant in the measurement of insulin deficient states of catabolism in patients with diabetes. A previous study of exhaled isoprene was found to be elevated during hypoglycemia. This study aims to expand on this to characterize the full range of changes in concentrations of volatile organic compounds in human breath during glucose fluctuations.

Characterizing this "biochemical fingerprint" of hypoglycemia may provide clues about what so-called diabetes alert dogs are detecting as well as improve our understanding of hypoglycemia, the physiology behind hypoglycemia unawareness, and potentially identify a novel non-invasive measure of blood glucose.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of type 1 diabetes
* No current or planned tobacco/nicotine use including vaping during the study
* Are not pregnant or planning to become pregnant during the study timeframe

Exclusion Criteria:

-

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with type 1 diabetes between age 5-80.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Absolute and relative change in concentration of measured volatile organic compounds in human breath in subjects with type 1 diabetes during hypoglycemia compared to euglycemia measured by proton-transfer-reaction time-of-flight mass spectrometry. | Until three low blood sugar events have occured with breath samples collected during low blood sugar and upon recovery to normal blood sugar; expected 1-2 weeks but allowed up to 1 month to complete sample collection
  Detectable difference in volatile organic compounds (anticipate up to 120-150 different ion signals to be assessed) in human breath during low blood sugar (<70 mg/dL) compared to normal blood sugar (70-180). As this is a 'hypothesis generating' pilot study, the investigators are observing what compounds are present and in what concentrations -- this is the reason for nonspecific outcome measures

SECONDARY OUTCOMES:
Characterize relationship of concentration of all measurable VOCs (anticipate 120-150 ion signals) by proton-transfer-reaction time-of-flight mass spectrometry across the spectrum of glycemia. | up to 1 month
  Statistically-significant (P<0.05) differences in concentration of volatile organic compounds in human breath in subjects with type 1 diabetes across the spectrum of glycemia (very low <54 mg/dL), low (55-69), in target (70-180), high (181-250), very high(>250))
Identify differences in patterns of exhaled VOCs in people who have hypoglycemia unawareness | up to 1 month
  Statistically significant (P<0.05) differences in patterns of exhaled VOCs between subjects with and without hypoglycemia unawareness identified by standardized hypoglycemia unawareness survey tools

CONTACTS AND LOCATIONS:
Overall Officials: Evan Los, MD, Principal Investigator — East Tennessee State Univerisity
Locations (1):
- Mountain States Health Alliance, Johnson City, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No